CLINICAL TRIAL: NCT06195085
Title: Long-term Outcomes of CT-guided Radioactive Iodine-125 Seed Implantation for Recurrent Desmoid Tumors
Brief Title: CT-guided Radioactive Iodine-125 Seed Implantation for Recurrent Desmoid Tumors
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: First Affiliated Hospital of the Army Medical University (Unknown); Shengli Oilfield Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RID
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Brachytherapy; Desmoid Tumor; Radioactive Iodine-125 Seed Implantation
MeSH Terms: conditions — Desmoid Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT-guided radioactive iodine-125 seed implantation: The patients, diagnosed with recurrent desmoid tumor, undergoing CT-guided radioactive iodine-125 seed implantation in 3 different centers including Peking University Third Hospital, First Affiliated Hospital of the Army Medical University, and Shengli Oilfield Central Hospital from July 2013 to July 2021.
  Interventions: Radiation: CT-guided radioactive iodine-125 seed implantation

INTERVENTIONS:
Radiation: CT-guided radioactive iodine-125 seed implantation — The CT-guided radioactive iodine-125 seed implantation procedure mainly consisted of preoperative treatment planning, intraoperative seed implantation and postoperative dosimetric evaluation. All procedures were performed as per relevant guidelines and regulations.

SUMMARY:
This study aimed to explore the long-term outcomes of CT-guided radioactive iodine-125 (I-125) seed implantation (RISI) for recurrent desmoid tumor.

A multicenter retrospective study reviewed 38 recurrent desmoid tumor patients receiving RISI from July 2013 to July 2021.The clinical outcomes including overall response rate (ORR), disease control rate (DCR), local control time (LCT), overall survival (OS), adverse events (AEs), and symptom relief rate were statistically assessed.

DETAILED DESCRIPTION:
Desmoid tumor was characterized by a high potential of recurrence even following initial definitive treatment. There were considerable controversies regarding the management of recurrent desmoid tumor. This study aimed to explore the long-term outcomes of CT-guided radioactive iodine-125 (I-125) seed implantation (RISI) for recurrent desmoid tumor.

38 patients, diagnosed with recurrent desmoid tumor, undergoing RISI in 3 different centers including Peking University Third Hospital, First Affiliated Hospital of the Army Medical University, and Shengli Oilfield Central Hospital from July 2013 to July 2021 were reviewed consecutively.

The clinical outcomes including overall response rate (ORR), disease control rate (DCR), local control time (LCT), overall survival (OS), adverse events (AEs), and symptom relief rate were statistically assessed.

ELIGIBILITY:
Inclusion Criteria:

1) recurrent desmoid tumor confirmed by pathologic or imaging diagnosis; 2) disease size ≥1 cm and ≤ 10 cm; 3) medically inoperable or individual refusal to resection; 4) Karnofsky performance status (KPS) ≥ 60; 5) adequate hematological reserves, hepatic function, renal function and heart function; 7) expected survival > 3 months.

Exclusion Criteria:

1) unconfirmed mass; 2) tumor invading the skin or mucous membrane; 2) patients with severe bleeding tendency; 3) patients with active infectious disease, trauma and severe wounds; 4) patients with any mental disorder; 5) patients with other somatic comorbidities of clinical concern; 6) pregnancy and lactation

Ages: 13 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patients, diagnosed with recurrent desmoid tumor, undergoing RISI in 3 different centers including Peking University Third Hospital, First Affiliated Hospital of the Army Medical University, and Shengli Oilfield Central Hospital from July 2013 to July 2021 were reviewed consecutively.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Local control time (LCT) | 8 years
  LCT was defined as the time from seed implantation to local progression
objective response rate (ORR) | 6 months
  ORR was calculated from patients achieving CR and PR
disease control rate (DCR) | 6 months
  DCR was likewise calculated from the patients of CR, PR and SD.

SECONDARY OUTCOMES:
overall survival (OS) | 8 years
  OS was defined as the time from RISI to death from any cause
adverse events (AEs) | 8 years
  The AEs were evaluated as per Radiation Therapy Oncology Group (RTOG) guidelines.
symptom relief rate | 8 years
  symptom relief rate was calculated from the patients achieving relief after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Always